CLINICAL TRIAL: NCT07186647
Title: Laparoscopic-Assisted Transanal Pull-Through for Hirschsprung Disease in Pediatric:Short and Intermediate Outcomes of Two Different Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelmaboud, assistant professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ped. -Surg.-77MED.-Research-00
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung Disease; Laparoscopy; Swenson; Soave; Pediatrics
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Intervention Model Description: A prospective, randomized study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 20 patients with HD
  Interventions: Procedure: laparoscopic-assisted Swenson-like (LASwL)
- Group B (Active Comparator): 20 patients with HD
  Interventions: Procedure: laparoscopic-assisted Soave (LASo)

INTERVENTIONS:
Procedure: laparoscopic-assisted Swenson-like (LASwL) — Following port placement, laparoscopic exploration was performed to evaluate the spastic colonic segment and transitional zone. An aperture was created in the sigmoid mesentery, and the sigmoid colon was mobilized. The proximal ganglionic bowel was mobilized while preserving the marginal arcades. The peritoneal reflection was sharply incised to facilitate dissection and mobilization of the aganglionic rectum. The procedure diverged between the two groups at this juncture: LASwl group: The rectum below the peritoneal reflection was dissected circumferentially up to a level 2 cm above the anal verge . LASo group: The rectum below the peritoneal reflection was minimally mobilized (within 1 cm of the peritoneal reflection). Following laparoscopic dissection, the ports were left in situ, and the position was adjusted for transanal dissection of the remaining rectum.
  Arms: Group A
Procedure: laparoscopic-assisted Soave (LASo) — Transanal endorectal procedure was conducted according to the standard technique described by De la Torre-Mondragon and Ortega-Salgado [12]. A circular incision was made in the mucosa, and mucosectomy was performed. The muscle sleeve was cut, connecting the two dissection planes circularly . After keeping the muscular cuff as short as possible, a longitudinal incision was made posteriorly. Then, the bowel was extracted, and the anastomosis was performed as described above.
  Arms: Group B

SUMMARY:
Compare the functional and surgical outcomes of laparoscopic-assisted Swenson-like (LASwL) and laparoscopic-assisted Soave (LASo) pull through in children with HD.

DETAILED DESCRIPTION:
A prospective, randomized study was conducted involving 80 patients diagnosed with HD at Al-Azhar University Hospitals over a 48-month period from September 2020 to August 2024. Participants were randomly allocated to the LASwL (Group A) or LASo (Group B). The primary outcome was the postoperative bowel function score. Secondary outcomes included operative time, blood loss, duration of hospital stay, and incidence of postoperative Hirschsprung-associated enterocolitis (HAEC).

ELIGIBILITY:
Inclusion Criteria:

* infants and children diagnosed with Hirschsprung's disease (HD) at the Department of Pediatric Surgery, Al-Azhar University Hospitals, from September 2020 to August 2024

Exclusion Criteria:

* Patients with ultrashort or total colonic aganglionosis and those who had previously undergone pull-through procedures

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative bowel function score | 2 years
  This assessment evaluated the ability to hold back defecation, the ability to feel or report the urge to defecate, the frequency of defecation, soiling accidents, constipation, and social issues. Most items are scored on a 0-3 scale, while defecation frequency is scored 1-2, resulting in a maximum total score of 20. A higher score indicates better bowel function, with Scores ranged from 17-20 (excellent), 12-16 (good), 9-11 (fair), and less than 8 (poor)

CONTACTS AND LOCATIONS:
Locations (1):
- pediatric surgery departments- Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided